CLINICAL TRIAL: NCT04222543
Title: Imaging of Tumour Microenvironment in Patients With Oropharyngeal Head and Neck Squamous Cell Carcinoma Using RGD PET/CT Imaging
Acronym: PIVOT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL69928.091.19
Record Dates: First submitted 2019-11-20; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-11

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: Tumour microenvironment; Chemoradiotherapy; Oropharyngeal squamous cell carcinoma; Human papilloma virus; Positron emission tomography
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cytidine Triphosphate

STUDY DESIGN:
Intervention Model Description: Imaging results of HPV positive tumours are compared to imaging results of HPV negative tumours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Negative tumours (Active Comparator): Patients will receive four scans.
  Interventions: Combination Product: RGD PET/CT
- HPV positive tumours (Active Comparator): Patients will receive four scans.
  Interventions: Combination Product: RGD PET/CT

INTERVENTIONS:
Combination Product: RGD PET/CT — Patients will receive an RGD PET/CT and a CT perfusion scan prior to treatment and during chemoradiotherapy
  Other Names: CT perfusion

SUMMARY:
Known risk factors inducing squamous cell carcinomas of the head and neck are tabacco and alcohol intake. However, the incidence of human papillomavirus (HPV) related oropharyngeal carcinomas is increasing. It is known that HPV+ and HPV- tumors have a different reaction to (chemo)radiotherapy. The exact mechanisms underlying these differences is not yet known but might be caused by changes in vascularity. Therefore the vasculature is imaged with the help of a study specific Gallium-68-DOTA-(RGD)2 PET/CT scan and a CT perfusion scan.

DETAILED DESCRIPTION:
The incidence of Human Papilloma Virus positive (HPV+) oropharyngeal Head and Neck Squamous Cell Carcinoma (HNSCC) is rising and it has become evident that this type of cancer represents a subgroup of HNSCC that is characterized by a more favourable prognosis, mediated by a distinct tumour microenvironment, compared to patients with HPV negative (HPV-) tumours. However, the exact mechanisms underlying this improved treatment outcome and the potential role of the tumour microenvironment are not fully understood yet. Imaging of αvβ3 integrin expression will obtain more insight in the differences in tumour microenvironment between HPV+ and HPV- oropharyngeal HNSCC. CT perfusion provides additional characterisation of this tumour microenvironment. Therefore, these techniques may have the potential to predict response to treatment and might possibly steer treatment decisions in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Proven squamous cell carcinoma of the oropharynx
* p-16 immunohistochemistry analysis
* Tumour lesion of at least 1.0 cm in diameter
* Planned chemoradiotherapy as primary treatment
* Ability to provide written informed consent

Exclusion Criteria:

* Contra-indications for PET
* Contra-indications for administration of iodine-containing contrast agents
* Other serious illness that can affect the scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Differences in RGD-tracer uptake between HPV positive and negative tumours | 1 month
  standardized uptake values (SUV) of Ga68-RGD
Differences in RGD-tracer uptake between the pre- and per-treatment scan | 1 month
  standardized uptake values (SUV) of Ga68-RGD
Differences in CT perfusion flow parameters between HPV positive and negative tumours | 1 month
  Determining the blood flow using ROIs of the tumour drawn on the contrast enhanced CT
Differences in CT perfusion parameters between HPV positive and negative tumours | 1 month
  Determining the blood volume using ROIs of the tumour drawn on the contrast enhanced CT
Differences in CT perfusion flow parameters between the pre- and per-treatment scan | 1 month
  Determining the blood flow using ROIs of the tumour drawn on the contrast enhanced CT
Differences in CT perfusion parameters between the pre- and per-treatment scan | 1 month
  Determining the blood volume using ROIs of the tumour drawn on the contrast enhanced CT

SECONDARY OUTCOMES:
Differences in RGD-tracer uptake between patients with locoregional control or recurrence within one year | 1 year
  standardized uptake values (SUV) of Ga68-RGD
Differences in CT perfusion flow parameters between patients with locoregional control or recurrence within one year | 1 year
  Determining the blood flow using ROIs of the tumour drawn on the contrast enhanced CT
Differences in CT perfusion parameters between patients with locoregional control or recurrence within one year | 1 year
  Determining the blood volume using ROIs of the tumour drawn on the contrast enhanced CT

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No